CLINICAL TRIAL: NCT05317481
Title: Reducing Suicide Risk in Adolescents and Young Adults Via a Psychobehavioral Intervention to Regularize Daily Rhythms and Improve Brain Circuitry Functioning
Brief Title: Reducing Suicide Risk in Adolescents and Young Adults Via a Psychobehavioral Intervention to Regularize Daily Rhythms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000032361; STR-1-002-20 (Other Grant/Funding Number: American Foundation for Suicide Prevention)
Record Dates: First submitted 2022-03-23; First posted 2022-04-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Bipolar Disorder; Major Depressive Disorder; Mood Disorders; Suicide; Suicidal Ideation
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Mood Disorders; Suicide; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: This is a randomized control trial (RCT) with subjects randomized 2:1 (using block randomization) to BE-SMART-DR or a psychoeducational control comparator condition (CC).
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BE-SMART-DR (Experimental): Participation will include research clinical/behavioral interviews and symptom self-ratings, magnetic resonance imaging (MRI) scanning, actigraphy wearables, and use of smart phones for ecological momentary assessment (EMA). Subjects will participate in 12 weekly sessions and 6-month in person follow-up.
  Interventions: Behavioral: BE-SMART-DR
- control comparator condition (Active Comparator): Matched for experimental, participation will include research clinical/behavioral interviews and symptom self-ratings, magnetic resonance imaging (MRI) scanning, actigraphy wearables, and use of smart phones for ecological momentary assessment (EMA). Subjects will participate in 12 weekly sessions and 6-month in person follow-up.
  Interventions: Behavioral: psychoeducational control comparator condition (CC)

INTERVENTIONS:
Behavioral: BE-SMART-DR — Therapy that provides self-directed strategies to regularize sleep and other DRs to reduce short-term suicide risk that can be used lifelong to potentially also reduce long-term suicide risk
  Arms: BE-SMART-DR
Behavioral: psychoeducational control comparator condition (CC) — Structured sessions, matched for BE-SMART-DR session number and time, that will emphasize established strategies to manage health and well being
  Arms: control comparator condition

SUMMARY:
The purpose of this study is to advance a non-pharmacologic suicide preventive intervention with wide dissemination potential as an innovative high-yield solution to reduce suicide rates. The investigators aim to achieve this with this study of Brain Emotion Circuitry Self-Monitoring and Regulation Therapy for Daily Rhythms (BE-SMART-DR), that provides self-directed strategies to regularize sleep and other DRs to reduce short-term suicide risk that can be used lifelong to potentially also reduce long-term suicide risk.

DETAILED DESCRIPTION:
This is a randomized control trial (RCT) with subjects randomized 2:1 (using block randomization) to BE-SMART-DR or a psychoeducational control comparator condition (CC). Participation will include research clinical/behavioral interviews and symptom self-ratings, magnetic resonance imaging (MRI) scanning, actigraphy wearables, and use of smart phones for ecological momentary assessment (EMA). Subjects will participate in 12 weekly sessions and 6-month in person follow-up.

Objectives

1. Show pre-post BE-SMART-DR suicidal ideation and propensity (SI/P) decreases associated with DR regularity and quality increases
2. Show pre-post BE-SMART-DR improvements in the functioning of a brain system that subserves emotional and other behavioral control (i.e., a hypothalamus-amygdala-ventral prefrontal cortex (vPFC), (HAV), system)

ELIGIBILITY:
Inclusion Criteria:

* with Diagnostic and Statistical Manual 5 (DSM5) Bipolar Disorder (BD) I, II or Otherwise Specified (OS) or Major Depressive Disorder (MDD)
* have a history of 1 or more suicide attempts and/or a score of at least 3 on the SSI

Exclusion Criteria:

* Significant medical or neurologic illness (especially if related to cerebral tissue)
* MRI contraindication,
* pregnancy by urine test
* current moderate or severe alcohol/other substance use disorders except caffeine/nicotine
* positive urine screen for benzodiazepines, cocaine, amphetamines, phencyclidine, opiates, oxycodone; not cannabis as its use is common in this population and it can remain positive for a month
* current evidence-based individual psychotherapy (e.g. cognitive behavioral therapy, dialectical behavioral therapy,) or treatment directly targeting brain regions of interest e.g. transcranial magnetic stimulation or electro-convulsive therapy,
* current psychosis
* inability to provide informed consent, including IQ<70, Young Mania Rating Scale (YMRS) >25, or too symptomatic by PI's judgment
* active suicidal plan or intent or Columbia Suicide Severity Rating Scale (C-SSRS) stage "4" risk (some intent to carry out the plan; as indicated by multisite study assessing suicide risk in randomized clinical trials or if revealed on any rating scale or in judgment of any study clinician.
* homicidal ideation

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Change in the experimental group from baseline in BE-SMART-DR Suicidal Ideation/Propensity (SI/P) using Beck Scale for Suicide Ideation (SSI) and Concise Health Risk Tracking Scale (CHRT) | baseline, during the intervention, immediately after the intervention
  Change in the experimental group from baseline in BE-SMART-DR Suicidal Ideation/Propensity (SI/P) using the interviewer assessed Beck Scale for Suicide Ideation (SSI), one of the most widely used measures to assess suicidal ideation. This is a 19 item scale with scores ranging from 0 to 38, with higher values indicating a greater risk of suicide. We will also use the Concise Health Risk Tracking Scale (CHRT), a brief self report measure. The CHRT Propensity score (9 items) covers the domains of pessimism, helplessness, despair and perceived lack of social support. Items are scored on a five-point Likert scale with responses ranging from "strongly disagree" (zero) to "strongly agree" (four), thereby creating a total propensity score that ranges from 0-36, with higher scores showing higher levels of suicidal propensity and suicidal thoughts.
Change from baseline in BE-SMART-DRs Daily Rhythms (DR) using the Brief Social Rhythm Scale (BSRS) | baseline, during the intervention, immediately after the intervention
  Change from baseline in BE-SMART-DRs Daily Rhythms (DR) will be assessed using the Brief Social Rhythm Scale (BSRS). This is a measure of DR regularity for 10 activities that include social contexts. It uses a scale ranging from 1 (very regularly) to 6 (very irregularly), with high mean scores indicating high irregularity. Summary scores are the average across all 10 items with higher scores indicating higher irregularity.
Change from baseline in BE-SMART-DRs Daily Rhythms (DR) using the Pittsburgh Sleep Quality Index (PSQI) | baseline, during the intervention, immediately after the intervention
  Change from baseline in BE-SMART-DRs Daily Rhythms (DR) using the Pittsburgh Sleep Quality Index (PSQI), a self-reported survey. The 10 items in the PSQI relate to usual sleep habits over the last month, including time it takes to fall asleep, usual bedtime, hours of sleep per night, as well as questions about the frequency of sleep issues (not during the past month, less than once per week, once or twice per week, or three or more times per week). Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Blumberg, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Magnetic Resonance Research Center, New Haven, Connecticut
  - Mood Disorders Research Program, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No